CLINICAL TRIAL: NCT06901401
Title: Oral Health-Related Quality of Life Using EORTC QLQ-H&N35 in Head and Neck Cancer Survivors Within the First Year Following Treatment: a Cross-Sectional Study in Egypt
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Other Study IDs: HAM00213
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cncer
Keywords: Oral Health-Related Quality of Life (OHRQoL); Head and Neck Cancer (HNC); EORTC QLQ-H&N35
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HNC Survivors' Oral Health and Quality of Life in Egypt: This cohort includes head and neck cancer (HNC) survivors within the first year post-treatment at Ahmed Maher Teaching Hospital (AMTH) in Egypt. The study evaluates Oral Health-Related Quality of Life (OHRQoL) using the EORTC QLQ-H&N35 questionnaire, along with clinical assessments like the Oral Hygiene Index-Simplified (OHI-S) and the WHO Oral Mucositis Scale.
  The research examines the impact of sociodemographic factors, oral hygiene practices, and treatment-related variables on oral health and overall quality of life, with a focus on radiotherapy and chemotherapy effects. While no interventions are applied, findings will support future strategies to improve post-treatment oral care for HNC survivors in Egypt.

SUMMARY:
This study aims to evaluate Oral Health-Related Quality of Life (OHRQoL) in head and neck cancer (HNC) survivors within the first year following treatment in Egypt. Using a cross-sectional study design, data will be collected from patients at Ahmed Maher Teaching Hospital (AMTH) through structured questionnaires and clinical assessments, including the Arabic version of EORTC QLQ-H&N35, oral hygiene index-simplified (OHI-S), and the WHO Oral Mucositis Scale.

The study will examine the association between OHRQoL and various factors, including sociodemographic characteristics, oral hygiene practices, and clinical parameters such as oral mucositis severity. A sample size of 112 participants was determined using a one-sample t-test, ensuring adequate statistical power while accounting for a 20% dropout rate.

Findings from this research will help highlight the impact of HNC treatment on oral health and provide insights into improving oral care strategies for better patient quality of life in Egypt.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the seventh most common cancer globally, accounting for more than 660,000 new cases and 325,000 deaths annually. The number of HNC cases is expected to grow by 30% each year until 2030.[1] The rise has been observed in both developed and developing countries.[2] The survival for HNC has improved modestly over the past three decades with the introduction of different and multi-disciplinary treatment modalities.[3] There are several treatment options for HNC, including radiation therapy, surgery, and chemotherapy. These treatments can be used alone or in combination. Radiation therapy (RT) involves using high-energy beams to destroy cancer cells, while it is an important part of HNC treatment, it can also cause various toxicities, sometimes severe, toxicities.[4].

In most of the cases, head and neck tumors may destroy organs that play an important part in daily activities such as eating and speaking [5]. Additionally, the therapeutic approaches for the treatment of cancer usually result in collateral effects [6]. that impact in the quality of life. The assessment of the quality of life in patients with cancer became a valuable tool to investigate the progression of the disease and the effectiveness of the treatment [7].

The oral condition has an essential role in the individual's systemic health [8]. In specific, the quality of lifer elated to oral health (OHRQoL) may be defined as the lack of negative impact of the oral condition on social, psychological and functional activities [9]. In general, patients with tumors in the oral cavity figure amongst the worst indices for the quality of life when compared to patients with tumors in other regions [10]. Based on the exposed, the present study aimed to measure the impact of OHRQoL of patients with HNC and to evaluate the factors associated.

QoL assessment is an important tool for evaluating not only the impact of disease and its treatment on an individual level but also helpful in developing and revising the rehabilitative ser- vices and patient education material to further improve the clinical outcomes (survival) of patients [11]. Oral health related quality of life (OHRQoL), specifically focuses on self-report aspects pertaining to oral health, capturing the functional, social, and psychological dimensions affected by oral disease [12]. In the case of HNC, disruptions in key oral functions poses a higher risk of adversely affecting both OHRQoL and overall QoL[13].

Not much evidence is found in Egypt related to oral care measures for HNC patients, such as professional care by a dentist and dental hygienist (mechanical or manual removal of mucosal debris, oral hygiene counsel- ling, etc.) at least once a week until the completion of RT [14]. The patients are often unaware of the potential harm from the cancer treatment, only a proportion of HNC patients seek dental consultation for their complications, and most of them suffer greatly even after the completion of treatment due to disturbed oral functions.

To the best of our knowledge, this study represents the first comprehensive assessment of OHRQoL in HNC treated patients who had completed their cancer treatment within the past 12 months. Additionally, it aims to explore the associations between various oral clinical parameters, including oral hygiene status and oral mucositis, and several predictive factors such as sociodemographic characteristics and treatment-related variables in relation to OHRQoL. The findings of this study will highlights the importance of standardizing oral care and improving oral health support for HNC treated patients to reduce the impact of oral problems which can negatively impact their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

(HNC).

* Completed cancer treatment (surgery, radiotherapy, and/or chemotherapy) within the past 12 months.
* Attending routine follow-up visits at Ahmed Maher Teaching Hospital (AMTH), Egypt.
* Able to communicate and complete the EORTC QLQ-H&N35 questionnaire.
* Presence of at least one molar and one central incisor in both upper and lower dentition (for oral hygiene assessment).
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Patients with cognitive impairment or severe mental illness affecting their ability to respond to the questionnaire.
* Patients with debilitating conditions (e.g., terminal illness, bedridden status).
* Trismus (mouth opening <20mm) preventing oral examination.
* Patients who decline to participate or withdraw consent.
* Patients with incomplete medical records or loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult head and neck cancer (HNC) survivors who have completed surgery, radiotherapy, and/or chemotherapy within the past 12 months. Participants will be recruited from the oncology unit at Ahmed Maher Teaching Hospital (AMTH) in Egypt during their routine follow-up visits.
  The study population will consist of individuals aged 18 years and older, representing diverse sociodemographic backgrounds. Eligibility criteria include patients who can communicate and complete the EORTC QLQ-H&N35 questionnaire, as well as those with at least one molar and one central incisor in both upper and lower dentition for oral hygiene assessment. Patients with cognitive impairments, severe debilitating conditions, or trismus (mouth opening <20mm) will be excluded.
  This study aims to evaluate the impact of cancer treatment on oral health-related quality of life (OHRQoL) and identify factors affecting post-treatment oral health outcomes in Egyptian HNC survivors.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Oral Health-Related Quality of Life (OHRQoL) Score | single point "Baseline"
  The Oral Health-Related Quality of Life (OHRQoL) Score will be assessed using the EORTC QLQ-H&N35 questionnaire, a validated tool for evaluating the impact of head and neck cancer (HNC) and its treatment on patients' oral health and overall quality of life. This questionnaire captures functional, social, and psychological aspects related to oral health, including pain, swallowing difficulties, dry mouth, speech problems, and social interactions.
  Scores range from 0 to 100, with higher scores indicating worse OHRQoL and greater impairment in daily activities. This measure will help identify factors influencing post-treatment oral health outcomes and guide future supportive care strategies for HNC survivors in Egypt

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Teaching Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided